CLINICAL TRIAL: NCT02993237
Title: A Study to Assess the Acceptability/Swallowability of DRV-containing FDC Tablets in HIV-1 Infected Adolescents, Using Matching Placebo Tablets
Brief Title: Study to Assess the Acceptability/Swallowability of DRV-Containing FDC Tablets in HIV-1 Infected Adolescents, Using Matching Placebo Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR108265; TMC114FD2HTX1003 (Other: Janssen Research & Development, LLC); 2016-003016-12 (EudraCT Number)
Record Dates: First submitted 2016-12-13; First posted 2016-12-15 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: HIV-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: DRV/COBI Placebo followed by D/C/F/TAF Placebo (Experimental): Participants will receive fixed dose combination (FDC) of darunavir/cobicistat (DRV/COBI) matching placebo tablets (Intake 1) and FDC of darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF) matching placebo tablets (Intake 2) on Day 1. Both the intakes will be separated by at least 30 minutes.
  Interventions: Drug: DRV/COBI FDC placebo tablet; Drug: D/C/F/TAF FDC placebo tablets
- Group 2: D/C/F/TAF Placebo followed by DRV/COBI Placebo (Experimental): Participants will receive FDC of D/C/F/TAF matching placebo tablets (Intake 1) and FDC of DRV/COBI matching placebo tablets (Intake 2) on Day 1. Both the intakes will be separated by at least 30 minutes.
  Interventions: Drug: DRV/COBI FDC placebo tablet; Drug: D/C/F/TAF FDC placebo tablets

INTERVENTIONS:
Drug: DRV/COBI FDC placebo tablet — Participants will receive 1 placebo tablet matching the DRV/COBI 800/150 milligram (mg) FDC
Drug: D/C/F/TAF FDC placebo tablets — Participants will receive 1 placebo tablet matching the D/C/F/TAF 800/150/200/10 mg FDC.

SUMMARY:
The primary purpose of this study is to assess the acceptability of swallowing the darunavir/cobicistat (DRV/COBI) and darunavir/cobicistat/emtricitabine/tenofovir alafenamide (D/C/F/TAF) fixed-dose combination (FDC) tablets, using matching placebo tablets, in human immunodeficiency virus (HIV) -1 infected adolescent patients.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be male or female between 12 to 17 years of age, inclusive
* Participant must have a body weight of at least 40 kilogram (kg)
* Informed consent must be obtained (from participant and/or his/her parent(s)/legal guardian, as applicable) and an age-appropriate Assent Form, as applicable, indicating that the purpose of, and procedures required for, the study are understood and that the participant is willing to participate in the study
* Participant must be able to comply with the protocol requirements, and adhere to prohibitions and restrictions specified in the protocol
* Participant has documented chronic human immunodeficiency virus (HIV) -1 infection, and is aware of his/her HIV-1 diagnosis
* Participant must be on a stable antiretroviral (ARV) regimen for at least 3 months and has documented plasma HIV-1 ribonucleic acid (RNA) less than (<) 50 copies/ milliLitre (mL) within 3 months prior to screening
* Participant must be willing to assess swallowability of the placebo tablets and be able to do so (as demonstrated by the intake of a reference placebo tablet)

Exclusion Criteria:

* Participant has any condition that, in the opinion of the Investigator, would compromise the study or the well-being of the participant, or prevent the participant from meeting or performing study requirements
* Participant has any condition that, in the opinion of the Investigator, could prevent, limit, or confound the protocol-specified assessments
* Participant has any active clinically significant physical or psychological disease or findings during screening that, in the Investigator's opinion, would compromise the participant's safety, ability to swallow (eg, candidiasis), or outcome of the study
* Participant has history of difficulty with oral intake of ARV therapy or other medications
* Participant is taking disallowed concomitant medications or over-the-counter products
* Participant is a family member of an employee or Investigator of the study site or Participant is a family member of an employee of Johnson & Johnson

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Proportion of Acceptability of Swallowing Fixed-Dose Combination (FDC) Tablets in Human Immunodeficiency Virus (HIV)-1 Infected Adolescent Patients | Day 1
  Swallowability will be assessed based on a 7-point questionnaire indicating how difficult/easy it was to swallow the tablet, ranging from "very difficult" to "very easy". The acceptability proportion is obtained by a dichotomization of the acceptability/swallowability scale, i.e. 'slightly difficult' or worse versus 'neither difficult nor easy' or better.

SECONDARY OUTCOMES:
Acceptability of Daily Intake of the FDC Tablets, by HIV-1 Infected Adolescent Participants | Day 1
  Acceptability for long term daily use will be assessed based on a 3-point questionnaire, 'not acceptable', 'acceptable', or 'good to take'.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (4):
- United States (4):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Emory University, Atlanta, Georgia
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Health Science Center, Houston, Texas

REFERENCES:
- See also: A study to assess the acceptability/swallowability of DRV-containing FDC tablets in HIV-1 infected adolescents, using matching placebo tablets — https://www.clinicaltrialsregister.eu/ctr-search/trial/2016-003016-12/results